CLINICAL TRIAL: NCT02732860
Title: Prospective Evaluation of Freshly Implanted Cancers in Mice to Test Drug Response in Matching Host
Brief Title: Personalized Patient Derived Xenograft (pPDX) Modeling to Test Drug Response in Matching Host
Acronym: REFLECT
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REFLECT-001
Record Dates: First submitted 2016-02-10; First posted 2016-04-11 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer; Breast Cancer; Breast Neoplasms; Ovarian Cancer; Ovarian Neoplasm
Keywords: personalized patient-derived xenografts (pPDX); molecular profiling; epigenetic analysis; drug sensitivity testing; triple negative; metastatic; serous
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, formalin fixed paraffin embedded blocks, fresh tumor tissue, malignant effusion or ascites (if no tumor tissue available), archival tissue (if not enrolled in molecular profiling studies IMPACT/OCTANE)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Triple Negative Breast Cancer: Triple negative breast cancer patients with residual invasive disease following neoadjuvant chemotherapy (n= up to 15) or with newly diagnosed metastatic disease (n=up to 30).
  After the screening procedures confirms patient eligibility:
  * Molecular Profiling will be performed on clinical sample
  * pPDX generation for in vivo drug testing
  * In vitro organoid culture generation (if sufficient fresh tissue available)
  * Identifying an actionable genomic alteration and drug making a matched treatment therapy recommendation.
  Interventions: Other: Molecular Profiling & In Vivo drug testing in pPDX and organoid cultures
- Colorectal Cancer: Colorectal cancer patients with metastatic disease undergoing resection of liver metastases, or with lesions amenable to biopsy (n=up to 15).
  After the screening procedures confirms patient eligibility:
  * Molecular Profiling will be performed on clinical sample
  * pPDX generation for in vivo drug testing
  * In vitro organoid culture generation (if sufficient fresh tissue available)
  * Identifying an actionable genomic alteration and drug making a matched treatment therapy recommendation.
  Interventions: Other: Molecular Profiling & In Vivo drug testing in pPDX and organoid cultures
- High Grade Serous Ovarian Cancer: High grade serous ovarian cancer patients with recurrent disease with a life expectancy of at least 12 months (n=up to 15), or Stage III or IV with residual disease following neoadjuvant chemotherapy, or at risk of high recurrence (n=up to 15).
  After the screening procedures confirms patient eligibility:
  * Molecular Profiling will be performed on clinical sample
  * pPDX generation for in vivo drug testing
  * In vitro organoid culture generation (if sufficient fresh tissue available)
  * Identifying an actionable genomic alteration and drug making a matched treatment therapy recommendation.
  Interventions: Other: Molecular Profiling & In Vivo drug testing in pPDX and organoid cultures
- Other tumor types: Other selected tumor types at the discretion of the PI (n= up to 30)
  After the screening procedures confirms patient eligibility:
  * Molecular Profiling will be performed on clinical sample
  * pPDX generation for in vivo drug testing
  * In vitro organoid culture generation (if sufficient fresh tissue available)
  * Identifying an actionable genomic alteration and drug making a matched treatment therapy recommendation.
  Interventions: Other: Molecular Profiling & In Vivo drug testing in pPDX and organoid cultures

INTERVENTIONS:
Other: Molecular Profiling & In Vivo drug testing in pPDX and organoid cultures — Molecular profiling of host tumour sample and pPDX will be performed and analyzed by an expert panel. In vitro organoid culture generation may also be performed if sufficient fresh tissue is available. Matched treatment recommendation based on profiling and in vivo pPDX drug testing results will be made, if available. This recommendation will be communicated to the primary oncologist.

SUMMARY:
By obtaining clinical specimens from participants with triple negative breast cancer (TNBC), colorectal cancer (CRC), high grade serous ovarian cancer (HGSOC), and other select tumor types to establish and profile as freshly implanted tumors in mice, the aim of this study is to identify agents with predicted activity in the host patient while also potentially providing them with personalized cancer treatment options

DETAILED DESCRIPTION:
Personalized patient-derived xenografts (pPDX) are increasingly used as tools for drug development in pre-clinical settings, and have been shown to recapitulate the histology and behavior of the cancers from which they are derived. Although, they have been commonly used productively as pre-clinical disease models to study disease biology and drug response, they have not been used prospectively to inform clinical management. pPDX have been employed to inform clinical decision-making in small studies, which have shown high concordance between individual pPDX and patient responses to therapy. While encouraging, the role of this approach in breast, colorectal, ovarian, and other cancer populations and in the context of genomic drug matching strategies remains undefined. This has created an opportunity to evaluate the utility of pPDX as clinical predictors to direct the use of chemo- and targeted therapies in combination with comprehensive genomic and epigenetic analysis for patients with TNBC, CRC, HGSOC and other selected tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Patient diagnosis must be categorized as either (I) OR (II) OR (III) OR (IV):

   (I) Histologically confirmed Triple Negative Breast Cancer by Institutional and American Society of Clinical Oncology (ASCO)/Cancer of American Pathologists (CAP) guidelines, either:
   * Stage IV (metastatic) disease that has not been treated with systemic therapy in the metastatic setting or
   * Stage I to III (non-metastatic) with residual mass by clinical exam and/or breast imaging following anthracycline + taxane-containing neoadjuvant chemotherapy

   OR

   (II) Histologically-confirmed Stage IV colorectal cancer treated with ≤ 1 line of systemic therapy in the metastatic setting, either:
   * Undergoing surgical resection of liver metastases or
   * With metastatic lesions amenable to biopsy

   OR

   (III) Histologically-confirmed advanced High Grade Serous Ovarian Cancer, either:
   * Recurrent disease with a life expectancy of at least 12 months or
   * Stage III or IV with residual disease following neoadjuvant chemotherapy, or at risk of high recurrence

   OR

   (IV) Histologically confirmed solid tumor not meeting criteria for (I), (II) or (III) above, for which evaluation of investigational therapies is of particular interest or where clinical need exists, at the discretion of the PI
3. Disease amenable to biopsy or surgery for tissue procurement
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Willingness and ability of patient to provide signed voluntary informed consent.

Exclusion Criteria:

1. Clinically significant hepatic, renal, cardiac or other organ dysfunction likely to limit participation in clinical trials.
2. Known brain metastasis
3. Any condition that could interfere with a patient's ability to provide informed consent such as dementia or severe cognitive impairment.
4. Any contraindication to undergoing a biopsy procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with TNBC, CRC, HGSOC, or selected other tumour types, referred to, or being treated at Princess Margaret Cancer Centre.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-12; Primary Completion 2026-01-04 (Estimated); Study Completion 2026-01-04 (Estimated)

PRIMARY OUTCOMES:
Measure of drug sensitive pPDX to a panel of drugs as a predictor of clinical response in matched host | up to 5 years
  Sensitivity measured by tumor growth inhibition (>80%) or objective tumor response (regression) as per Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
Rate of results reporting | up to 5 years
Rate of pPDX engraftment | up to 2 years

SECONDARY OUTCOMES:
Comparison of actionable alterations identified in clinical and pPDX samples | up to 5 years
  Genomic alterations identified using the Ion Proton System for Next-Generation Sequencing (NGS).
Number of patients with molecular abnormalities in pPDX as identified via NGS eliciting clinical responses while receiving matched treatments. | up to 5 years
  Overall accuracy of clinical responses as assessed by RECIST criteria in patient tumor.
Correlation between pPDX and organoid drug sensitivities | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Cescon, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada